CLINICAL TRIAL: NCT04344041
Title: COvid-19 and Vitamin D Supplementation: a Multicenter Randomized Controlled Trial of High Dose Versus Standard Dose Vitamin D3 in High-risk COVID-19 Patients (CoVitTrial)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Collaborators: Mylan Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-001602-34
Record Dates: First submitted 2020-04-09; First posted 2020-04-14 (Actual); Last update posted 2021-04-30 (Actual); Status verified 2021-04

CONDITIONS: Coronavirus
Keywords: vitamin D; older adults
MeSH Terms: conditions — Coronavirus Infections | interventions — Cholecalciferol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): High dose of vitamin D3
  Interventions: Drug: cholecalciferol 200,000 IU
- Comparator group (Active Comparator): Standard dose of vitamin D3
  Interventions: Drug: cholecalciferol 50,000 IU

INTERVENTIONS:
Drug: cholecalciferol 200,000 IU — Patients receive a vitamin D supplementation of 400,000 IU in a single oral dose.
  Arms: Intervention group
Drug: cholecalciferol 50,000 IU — Patients receive a vitamin D supplementation of 50,000 IU in a single oral dose
  Arms: Comparator group

SUMMARY:
Vitamin D is a secosteroid hormone produced by the skin during Summer exposure to UVB rays. Hypovitaminosis D is common in Winter (October to March) at Northern latitudes above 20 degrees North, and from April to September at Southern latitudes beyond 20 degrees below the equator.

In the past, coronaviruses and influenza viruses have exhibited very high seasonality, with outbreaks occurring preferentially during the Winter. The Covid-19 pandemic is indeed more severe above Winter latitudes of 20 degrees, while it remains until now less severe in the Southern hemisphere, with a much lower number of deaths.

Preclinical research suggests that the SARS-Cov-2 virus enters cells via the angiotensin converting enzyme 2 (ACE2). Coronavirus viral replication downregulates ACE2, thereby dysregulating the renin-angiotensin system (RAS) and leading to a cytokine storm in the host, causing acute respiratory distress syndrome (ARDS).

Research also shows that vitamin D plays a role in balancing RAS and in reducing lung damage. On the contrary, chronic hypovitaminosis D induces pulmonary fibrosis through activation of RAS. Similarly, hypovitaminosis D has been strongly associated in the literature with ARDS, as well as with a pejorative vital prognosis in resuscitation but also in geriatric units, and with various comorbidities associated to deaths during SARS-Cov-2 infections. Conversely, vitamin D supplementation has been reported to increase immunity and to reduce inflammatory responses and the risk of acute respiratory tract infections.

High-dose oral vitamin D3 supplementation has been shown to decrease short-term mortality in resuscitation patients with severe hypovitaminosis D (17% absolute risk reduction). It is considered safe to take oral vitamin D supplementation at doses up to 10,000 IU/day for short periods, particularly in older adults, i.e. a population that is mostly affected by hypovitaminosis D and who should receive at least 1,500 IU of vitamin D daily to ensure satisfactory vitamin D status.

Vitamin D supplementation is mentioned as a potentially interesting treatment for SARS-Cov-2 infection but on a scientific basis with a low level of evidence until now.

We hypothesize that high-dose vitamin D supplementation improves the prognosis of older patients diagnosed with COVID-19 compared to a standard dose of vitamin D.

DETAILED DESCRIPTION:
• Inclusion visit A clinical examination is carried out. Social-demographic measures, health history, clinical examination measures (including OSCI score) and biological measures are collected.

Randomization is conducted on the day of the inclusion visit. The ZYMAD® 400,000 IU (2 vials of 200,000 IU) or 50,000 IU (1 vial of 50,000 IU) treatment is given to the patient.

* Visit at day 7 A blood test is carried out by a nurse to determine the serum 25-OHD, creatrinine, albumine and calcium concentrations.
* Visit at day 14 A visit or telephone call allows recording the onset of clinical events of interest. The drugs received as part of the usual treatment during the last 14 days are collected.
* Visit at day 28 A visit or telephone call allows recording the onset of clinical events of interest. The drugs received as part of the usual treatment during the last 14 days are collected.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 65 years old
* Infection with COVID-19 diagnosed with RT-PCR SARS-CoV-2 or withCT-scan of the chest suggesting viral pneumonia of peripheral predominance in a clinically relevant context
* Patient seen in hospitalization or consultation or in nursing home
* Diagnosed within the preceding 3 days
* Having at least one of the following two risk factors for complications:

  * age ≥75 years
  * Peripheral capillary oxygen saturation (SpO2) ≤ 94% ambient air, or a partial oxygen pressure (PaO2) to fraction of inspired oxygen (FiO2) ratio ≤ 300 mmHg
* Patients affiliated with or benefitting from a social security scheme
* Written and signed consent of the patient or a relative or legal representative or, if not possible, emergency inclusion procedure

Exclusion Criteria:

* Organ failure requiring admission to a resuscitation or high dependency unit
* Comorbidity that is life-threatening in the short-term (life expectancy <3 months)
* Any reason that makes follow-up at day 28 impossible
* Vitamin D supplementation in the previous month, with the exception of treatment providing less than 800 IU of vitamin D per day
* Contraindication for vitamin D supplementation: active granulomatosis (sarcoidosis, tuberculosis, lymphoma), history of calcic lithiasis, known hypervitaminosis D or hypercalcemia, known intolerance to vitamin D
* Participation in another simultaneous trial
* Safeguard of justice
* Peripheral capillary oxygen saturation (SpO2) ≤92% in spite of an oxygen therapy > 5L/min

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 260 (Actual)
Dates: Start 2020-04-15 (Actual); Primary Completion 2021-01-14 (Actual); Study Completion 2021-01-14 (Actual)

PRIMARY OUTCOMES:
Number of death of any cause, during the 14 days following the inclusion and intervention. | Day 14

SECONDARY OUTCOMES:
Number of death of any cause, during the 28 days following the inclusion and intervention. | Day 28
Clinical evolution between day 0 and day 14 based on the change of the WHO Ordinal Scale for Clinical Improvement (OSCI) for COVID-19 | Day 14
  OSCI ranges from 0 to 8, higher score meaning poorer outcome
Clinical evolution between day 0 and day 28 based on the change of the OSCI for COVID-19 | Day 28
  OSCI ranges from 0 to 8, higher score meaning poorer outcome
Rate of patients with at least one severe adverse event at day 28, according to the regulations | Day 28
Number of death of any cause during the 14 days following the inclusion and intervention, in patients with severe hypovitaminosis D (25-OHD <25nmol/L) at baseline | Day 14
Number of death of any cause during the 28 days following the inclusion and intervention, in patients with severe hypovitaminosis D (25-OHD <25nmol/L) at baseline | Day 28
Clinical evolution between day 0 and day 14 based on the change of the OSCI for COVID-19, in patients with severe hypovitaminosis D (25-OHD <25nmol/L) at baseline | Day 14
  OSCI ranges from 0 to 8, higher score meaning poorer outcome
Clinical evolution between day 0 and day 28 based on the change of the OSCI for COVID-19, in patients with severe hypovitaminosis D (25-OHD<25nmol/L) at baseline | Day 28
  OSCI ranges from 0 to 8, higher score meaning poorer outcome
Number of death of any cause during the 14 days following the inclusion and intervention, depending on serum vitamin D concentration achieved at day 7 (25-OHD<75nmol/L or 25-OHD≥75nmol/L) | Day 14
Number of death of any cause during the 28 days following the inclusion and intervention, depending on serum vitamin D concentration achieved at day 7 (25-OHD<75nmol/L or 25-OHD≥75nmol/L) | Day 28
Clinical evolution between day 0 and day 14 based on the change of the OSCI for COVID-19, depending on serum vitamin D concentration achieved at day 7 (25-OHD<75nmol/L or 25-OHD≥75nmol/L) | Day 14
  OSCI ranges from 0 to 8, higher score meaning poorer outcome
Clinical evolution between day 0 and day 28 based on the change of the OSCI for COVID-19, depending on serum vitamin D concentration achieved at day 7 (25-OHD<75nmol/L or 25-OHD≥75nmol/L) | Day 28
  OSCI ranges from 0 to 8, higher score meaning poorer outcome
Number of death of any cause during the 14 days following the inclusion and intervention, in patients with severe hypovitaminosis D (25-OHD<25nmol/L) at day 0, depending on serum vitamin D concentration achieved at day 7 (<75nmol/L or ≥75nmol/L) | Day 14
Number of death of any cause during the 28 days following the inclusion and intervention, in patients with severe hypovitaminosis D (25-OHD<25nmol/L) at day 0, depending on serum vitamin D concentration achieved at day 7 (<75nmol/L or ≥75nmol/L) | Day 28
Clinical evolution between day 0 and day 14 based on the change of the OSCI for COVID-19, in patients with severe hypovitaminosis D (25-OHD<25nmol/L) at day 0, depending on serum vitamin D concentration achieved at day 7 (<75nmol/L or ≥75nmol/L) | Day 14
  OSCI ranges from 0 to 8, higher score meaning poorer outcome
Clinical evolution between day 0 and day 28 based on the change of the OSCI for COVID-19, in patients with severe hypovitaminosis D (25-OHD<25nmol/L) at day 0, depending on serum vitamin D concentration achieved at day 7 (<75nmol/L or ≥75nmol/L) | Day 28
  OSCI ranges from 0 to 8, higher score meaning poorer outcome
Number of death of any cause during the 14 days following the inclusion and intervention, depending on evolution of serum vitamin D concentration between day 0 and day 7 | Day 14
Number of death of any cause during the 28 days following the inclusion and intervention, depending on evolution of serum vitamin D concentration between day 0 and day 7 | Day 28
Clinical evolution between day 0 and day 14 based on the change of the OSCI for COVID-19, depending on evolution of serum vitamin D concentration between day 0 and day 7 | Day 14
  OSCI ranges from 0 to 8, higher score meaning poorer outcome
Clinical evolution between day 0 and day 28 based on the change of the OSCI for COVID-19, depending on evolution of serum vitamin D concentration between day 0 and day 7 | Day 28
  OSCI ranges from 0 to 8, higher score meaning poorer outcome
Number of death of any cause during the 14 days following the inclusion and intervention, compared to mortality data in French hospital geriatric units from the current national survey by the French Society of Geriatrics and Gerontology | Day 14

CONTACTS AND LOCATIONS:
Locations (9):
- France (9):
  - CHU Angers, Angers
  - CHU Bordeaux, Bordeaux
  - CH Le Mans, Le Mans
  - CHU Limoges, Limoges
  - CHU Nantes, Nantes
  - CHU Nice, Nice
  - CHU Saint Etienne, Saint-Etienne
  - CH Saumur, Saumur
  - CHU Tours, Tours

REFERENCES:
- [Derived] Annweiler C, Beaudenon M, Gautier J, Gonsard J, Boucher S, Chapelet G, Darsonval A, Fougere B, Guerin O, Houvet M, Menager P, Roubaud-Baudron C, Tchalla A, Souberbielle JC, Riou J, Parot-Schinkel E, Celarier T; COVIT-TRIAL study group. High-dose versus standard-dose vitamin D supplementation in older adults with COVID-19 (COVIT-TRIAL): A multicenter, open-label, randomized controlled superiority trial. PLoS Med. 2022 May 31;19(5):e1003999. doi: 10.1371/journal.pmed.1003999. eCollection 2022 May. PMID 35639792
- [Derived] Shakoor H, Feehan J, Al Dhaheri AS, Cheikh Ismail L, Ali HI, Alhebshi SH, Apostolopoulos V, Stojanovska L. Role of vitamin D supplementation in aging patients with COVID-19. Maturitas. 2021 Oct;152:63-65. doi: 10.1016/j.maturitas.2021.03.006. Epub 2021 Mar 16. No abstract available. PMID 33757717
- [Derived] Annweiler C, Beaudenon M, Gautier J, Simon R, Dubee V, Gonsard J, Parot-Schinkel E; COVIT-TRIAL study group. COvid-19 and high-dose VITamin D supplementation TRIAL in high-risk older patients (COVIT-TRIAL): study protocol for a randomized controlled trial. Trials. 2020 Dec 28;21(1):1031. doi: 10.1186/s13063-020-04928-5. PMID 33371905